CLINICAL TRIAL: NCT06216184
Title: Adding Vortexing to the Maki Technique Provides no Benefit
Brief Title: Adding Vortexing to the Maki Technique Provides no Benefit for the Diagnosis of Catheter-related Bacteremia
Status: Completed | Type: Observational
Sponsor: University Hospital of Canary Islands (Other)
Responsible Party: Principal Investigator, Leonardo Lorente, Medical assistant, University Hospital of Canary Islands
Other Study IDs: CHUC_2022_17
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Catheter-related Bloodstream Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRI: Patients with suspected catheter-related infection (CRI) and with one central venous catheter for at least 7 days were included. The area under the curve (AUC) of the Maki technique, the vortexing technique and the combination of both techniques for the diagnosis of catheter tip colonization (CTC) and diagnosis of catheter-related bloodstream infection (CRBSI) were compared.
  Interventions: Diagnostic Test: Vortexing

INTERVENTIONS:
Diagnostic Test: Vortexing — use combined of vortexing and Maki techniques

SUMMARY:
The investigators wanted to determine whether the combined use of vortexing and Maki techniques provides profitability versus the Maki technique for the diagnosis of catheter tip colonization and catheter-related bloodstream infection

DETAILED DESCRIPTION:
BACKGROUND A previous study compared vortexing and Maki techniques for the diagnosis of catheter-related bloodstream infection (CRBSI), and concluded that vortexing was not superior to Maki method.

AIM To determine whether the combined use of vortexing and Maki techniques provides profitability versus the Maki technique for the diagnosis of catheter tip colonization (CTC) and CRBSI.

METHODS Observational and prospective study carried out in an Intensive Care Unit. Patients with suspected catheter-related infection (CRI) and with one central venous catheter for at least 7 days were included. The area under the curve (AUC) of the Maki technique, the vortexing technique and the combination of both techniques for the diagnosis of CTC and CRBSI were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of catheter-related infection (CRI) and with long term CVC (at least 7 days)

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient recruitment was performed in the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
diagnosis of catheter related bloodstream infection | 6 months
  Number of patients with vortexing and/or Maki technique positive

CONTACTS AND LOCATIONS:
Locations (1):
- Leonardo Lorente, San Cristóbal de La Laguna, Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No
The study is completed